CLINICAL TRIAL: NCT03939559
Title: The Efficiency of Home Based Dual Task Training in Parkinson Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Burcu Ersoz Huseyinsinoglu, Assoc.Prof., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: İstanbulUCerrahpasa
Record Dates: First submitted 2019-05-03; First posted 2019-05-07 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Parkinson Disease
Keywords: dual task; balance; postural control; rehabilitation; home-based exercise
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Patients who meet the inclusion criteria of the study will be included in the study and will be randomized into two groups.
Who Masked: Outcomes Assessor
Masking Description: Home exercise training and assessments will be provided by different physiotherapists. The evaluator physiotherapist will be blind to the treatment group to which the patient belongs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance Exercises Group (Experimental): Balance exercises group, 4 exercise packages which include static, dynamic and functional balance exercises will be taught in the first part of exercise period for 4 weeks. After the four weeks, the exercises should be progressed in the last 4 weeks in the second training session
  Interventions: Procedure: Static, dynamic and functional balance exercises
- Dual Task Based Balance Exercises Group (Experimental): Dual task based balance exercises group, 4 exercise packages which include static, dynamic and functional balance exercises with cognitive or motor dual task will be taught in the first part of exercise period for 4 weeks.
  Interventions: Procedure: Static, dynamic and functional balance exercises with dual task

INTERVENTIONS:
Procedure: Static, dynamic and functional balance exercises — In the first group (G1), 4 exercise packages which include static, dynamic and functional balance exercises will be taught in the first part of exercise period for 4 weeks
  Arms: Balance Exercises Group
Procedure: Static, dynamic and functional balance exercises with dual task — In the second group (G2), 4 exercise packages which include static, dynamic and functional balance exercises with cognitive or motor dual task will be taught in the first part of exercise period for 4 weeks.
  Arms: Dual Task Based Balance Exercises Group

SUMMARY:
The aim of this study was to investigate the effects of dual task home based exercise program on balance, gait and cognitive functions. The study is planned to include 60 patients with Parkinson's disease, whose levels are 1-3 according to the Hoehn-Yahr scale and will be admitted to Istanbul University Capa Medical Faculty Neurology Department Movement and Behavior Disorders Unit between June 2019 and February 2020. The aim of the study, duration, possible side effects of treatment will be given to the volunteers to participate in the study. The "Informed Consent Form am prepared in accordance with the standards determined by the Clinical Research Ethics Committee of Istanbul Faculty of Medicine will be approved and the study will be conducted in accordance with the Declaration of Helsinki.

Patients who meet the inclusion criteria of the study will be included in the study and will be randomized into two groups. Both groups will be given information with brochures containing the importance of exercise in Parkinson's disease and will be given DVD copies with weekly recordings. The time and activity schedule created at the end of the brochures will be required to record daily home exercises of the patients. In the balance exercises group; static, dynamic and functional balance exercise packages will be taught in Parkinson 's disease. In the dual task based balance exercises group; motor or cognitive dual task training will be combined these static dynamic and functional balance exercises. In both groups, exercises will be performed 3 days a week for 8 weeks.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effects of dual task home based exercise program on balance, gait and cognitive functions. The study is planned to include 60 patients with Parkinson's disease, whose levels are 1-3 according to the Hoehn-Yahr scale and will be admitted to Istanbul University Capa Medical Faculty Neurology Department Movement and Behavior Disorders Unit between June 2019 and February 2020. The aim of the study, duration, possible side effects of treatment will be given to the volunteers to participate in the study. The "Informed Consent Form am prepared in accordance with the standards determined by the Clinical Research Ethics Committee of Istanbul Faculty of Medicine will be approved and the study will be conducted in accordance with the Declaration of Helsinki.

Patients who meet the inclusion criteria of the study will be included in the study and will be randomized into two groups. Both groups will be given information with brochures containing the importance of exercise in Parkinson's disease and DVD copies where the exercises are recorded weekly. The time and activity schedule created at the end of the brochures, daily recording of home exercises of the patients will be requested. Home exercise training and assessments will be provided by different physiotherapists. The evaluator physiotherapist will be blind to the treatment group to which the patient belongs. In the balance exercises group; 4 exercise packages which include static, dynamic and functional balance exercises will be taught in the first part of exercise period for 4 weeks. After the four weeks, the exercises should be progressed in the last 4 weeks in the second training session. In the dual task based balance exercises group; 4 exercise packages which include static, dynamic and functional balance exercises with cognitive or motor dual task will be taught in the first part of exercise period for 4 weeks. After the four weeks, the exercises should be progressed in the last 4 weeks in the second training session.

The number of subjects to be taken for each group in the 95% confidence interval was considered to be 26, considering the minimal clinical significant change (Minimal Clinically Important Difference, MCID) 3.5 for the Timed Up and Go Test. Considering that the patients did not continue treatment, it was decided to take 30 patients to each group and to carry out the study with a total of 60 patients. The primary outcomes are Mini Best Test,Timed Get Up and Go Test. Also objective datas will be obtained from Biodex Balance System, Wii Balance Board and G Walk Sensory Walking System.The secondary outcome measures include activity balance confidence scale, Parkinson's Disease Questionnaire-39 and cognitive tests such as number range test, verbal memory processes test, mental flexibility and word fluency test.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 1-3 levels according to Hoehn Yahr scale
* Have 3 or fewer scores in the Freezing of Gait Questionnaire
* Obtain at least 24 points from the Mini Mental State Assessment test
* Independent walking on a flat surface without an auxiliary device

Exclusion Criteria:

* Serious hearing or vision problems
* Have any cardiac or orthopedic disorder that may prevent walking be
* Any other neurological disorder (eg, dementia, cerebrovascular disease)
* To have a level of education of less than 5 years.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-10 (Estimated); Primary Completion 2019-09-10 (Estimated); Study Completion 2020-02-10 (Estimated)

PRIMARY OUTCOMES:
Mini Best Test | 8 weeks
  The Mini-BEST test to be used for dynamic balance assessment is a 14-item balance scale and is a one-dimensional and highly reliable measurement method that requires approximately 15 minutes to complete.
Wii Balance Board | 8 weeks
  With the Wii Balance Board (WDT), the patients' static balances will be evaluated.
  The WDT includes a component similar to a typical force platform with four strain gauge based load sensors that can obtain data about changes in the pressure center and can be wirelessly connected to a computer via Bluetooth.
Biodex Balance System | 8 weeks
  The Biodex Balance System (BBS; Biodex Medical System Inc., Shirley, NY, USA) will be used to measure the displacement of the foot pressure center (CoP).
Timed Up and Go Test | 8 weeks
  Timed Up and Go Test is a simple, widely used and rapid test for assessing mobility, balance and fall risk
Gait Assessment with G walk | 8 weeks
  Spatio temporal parameters of the gait are planned to be evaluated using the G-walk sensor.

SECONDARY OUTCOMES:
Activity Balance Confidence Scale | 8 weeks
  Activity-Specific Balance Confidence Scale will be used to measure patient's balance confidence. The ABC questionnaire, which is answered by an individual's self-perception of 16 items, measures the perceived ability of an individual on a 0-100 scale to achieve equilibrium under different conditions. This item is used to lead into each activity considered: "how confident are you that you will not lose your balance or become unsteady when you...". Each item is rated on a rating scale that ranges from 0-100. The highest score shows full confidence in the balance abilities. Overall score is calculated by adding item scores and then dividing by the total number of items.
Parkinson Disease Questionnaire- 39 | 8 weeks
  PDQ-39 is a self-report survey using the 5-point Likert scale to assess quality of life in Parkinson Disease. 39 multiple choice items covering 8 dimensions such as: mobility, activity of daily living (ADL), Emotional well-being, Stigma, Social Support, Cognition,Communication, Bodily Discomfort. All items are accepted to impact quality of life and must be answered to compute scores for each dimension. The responded items based on the experiences from the preceding month and 5 point ordinal scoring system (0:never, 1:occasionally, 2:sometimes, 3:often,4:always). Dimension scores are computed by the sum of scores of each item in the related dimension divided by the maximum possible score of all the items in the dimension, multiplied by 100. Each dimension total score range from 0(never difficulty) to 100(always difficulty) and. Highest scores reflect worse quality of life. Overall score is the sum of dimension total scores divided by 8.
Number Range Test | 8 weeks
  Number Range Test consists of two parts. The first part is the forward number range, the second part is the reverse number range. The two parts are applied separately. In both sections, the numbers are one by one. First, the advanced number range is applied. Then, the countdown range is applied. The numbers are read to the subject so that a number is read per second. In both the forward and backward range, the subject is passed to the next attempt at any successful attempt. If both attempts fail, the test is not continued. Creates a range of digits of the last repeatable sequence
Verbal Memory Processes Test | 8 weeks
  The Verbal Memory Processes Test can distinguish many memory related parameters. The first of these; the instant memory of the person; the process of learning or acquiring knowledge, the third; remembering and recalling and remembering processes.
Mental Flexibility Test | 8 weeks
  As part of the Mini-Mental State Assessment test, the output from 100 to 7 is done up to 65 (100, 93, 86, 79, 72, 65). Every correct transaction gets 1 point
Word Fluency Test | 8 weeks
  F, A or S starting with the letter of the word or non-action words in as much as possible to say is based on a minute. Each letter is given 1 minute. The total score is all the words spoken in all letters. Measures verbal-phonological fluency. In the investigator's country, K, A, S letters were used in the standardization study. In this study, the total number of words will be taken into consideration.

CONTACTS AND LOCATIONS:
Overall Officials: Guzin Kaya Aytutuldu, MSc., Study Chair — Yeditepe University; Yonca Zenginler Yazgan, Assist.Prof., Study Chair — Istanbul University - Cerrahpasa

IPD SHARING:
Plan to Share IPD: No